CLINICAL TRIAL: NCT04096482
Title: Safety and Effectiveness Evaluation of the Peregrine Drivable ENT Scope for Office Endoscopy of the Paranasal Sinuses in Patients Who Underwent ESS
Brief Title: Safety and Effectiveness of the Peregrine Drivable ENT Scope for Endoscopy of the Paranasal Sinuses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early findings identified the need to update the design of the study device.
Sponsor: Emory University (Other)
Collaborators: 3NT Medical Ltd. (Industry)
Responsible Party: Principal Investigator, Joshua M. Levy, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00110282
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Sinus Problem
Keywords: Nasal endoscopy
MeSH Terms: interventions — Endoscopes

STUDY DESIGN:
Intervention Model Description: Patients who have had prior ESS and are scheduled for nasal endoscopy as part of a routine post-operative office visit or due to recurrence of symptoms will be evaluated with the standard endoscope followed by the Peregrine Endoscope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Standard 30° 4mm Endoscope Followed by Peregrine Endoscope (Experimental): Participants will receive an endoscopy with the standard 30° 4mm endoscope followed by an endoscopy with the Peregrine Drivable ENT Scope.
  Interventions: Device: Peregrine Drivable ENT Scope; Device: Standard 30° 4mm Endoscope

INTERVENTIONS:
Device: Peregrine Drivable ENT Scope — Peregrine, developed by 3NT Medical, is a single-use disposable handheld endoscope, which is thinner and more flexible than other endoscopes. The endoscope includes a camera at its end and a working channel. The thin endoscope provides a means to visualize the nasal cavity and paranasal sinus space and to deliver irrigation to treat the sinus ostia (drainage openings) and spaces within the paranasal sinus cavities
Device: Standard 30° 4mm Endoscope — The Standard 30° 4mm endoscopic sinus evaluation is the standard procedure that would normally be used to evaluate the condition of each participant.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Peregrine endoscope in patients in the office setting in terms of access into and visualization of the paranasal sinus anatomy, image quality, patient tolerability and clinical utility. Up to 30 participants who have had prior endoscopic sinus surgery (ESS) and are scheduled for nasal endoscopy in the office as part of a routine post-operative office visit or due to recurrence of symptoms, will be evaluated with the Peregrine Endoscope as well as a standard endoscope. This study aims to:

* compare visualization success rates of the paranasal sinus anatomy by Peregrine and by a standard endoscope used in the office setting.
* examine device related adverse events.
* assess the adequacy of the image quality of Peregrine for endoscopy procedures in the office.
* evaluate patient tolerability and pain

DETAILED DESCRIPTION:
Nasal endoscopy is a minimally invasive, diagnostic medical procedure and currently the most preferred initial method of evaluating medical problems affecting nose and sinuses such as nasal stuffiness and obstruction, sinusitis, nasal polyposis, nasal tumors, epistaxis, recurrent bouts of sneezing and rhinorrhea. Overall, the procedure is considered very safe and low-risk. Currently, nasal endoscopy can be performed with a flexible or rigid endoscope, typically after a topical decongestant and anesthetic are applied to the nasal mucosa.

Reprocessing is an issue of concern, especially for flexible endoscopes where multiple steps were confirmed to be critical for reprocessing to be effective. High-level disinfection has been determined to be the minimum level of disinfection required, which involves multiple steps including manual cleaning, leak testing, cleaning with an enzymatic agent, high-level disinfection, and drying with vertical storage. 3NT Medical Ltd. has developed the Peregrine Drivable Ear Nose and Throat (ENT) Scope, which offers the convenience of a single-use endoscope component coupled with performance characteristics of commercially available state-of-the-art reusable endoscopy systems. The single-use endoscope essentially removes concerns related to burdensome reprocessing techniques of a delicate tool required to achieve high-level of its disinfection.

The objective of this study is to assess the safety and performance of the Peregrine endoscope in patients in the office setting in terms of access and visualization of the paranasal sinus anatomy, image quality, and patient tolerability and pain. For this study, up to 30 patients who have had prior endoscopic sinus surgery (ESS) and who are scheduled for nasal endoscopy in the office, as part of a routine post-operative office visit or due to recurrence of symptoms, will be evaluated with Peregrine Endoscope. Access and visualization by an additional standard endoscope will be conducted and compared to Peregrine endoscope. Image quality of the Peregrine endoscope, participant tolerability and pain, and the impact of Peregrine on clinical decision making will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* A male or female patient who has had prior ESS and who is indicated for office endoscopy by the ENT specialist
* A patient who is able to understand the requirements of the study, is willing to comply with its instructions and schedules, and agrees to sign the informed consent form

Exclusion Criteria:

* Any medical disorder which in the investigator's judgment contraindicates the patient's participation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Levy, MD, Principal Investigator — Emory University
Locations (1):
- Emory Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial and after deidentification will be available for sharing.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing immediately following the embargo period associated with publication.
Access Criteria: Data will be available for sharing with primary investigators at academic institutions for the purposes of meta-analysis or nested studies with agreed publication plan. Data can be requested by contacting the study team and completing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital Midtown in Atlanta, Georgia, USA. Participant enrollment began November, 5, 2019 and all follow up was complete by September 1, 2020.
Groups:
- Standard 30° 4mm Endoscope Followed by Peregrine Endoscope: Participants with prior endoscopic sinus surgery (EES) scheduled for nasal endoscopy who are receiving an endoscopy with the standard 30° 4mm endoscope followed by an endoscopy with the Peregrine Drivable Ear Nose and Throat (ENT) Scope.
Period: Overall Study
Arm/Group | Standard 30° 4mm Endoscope Followed by Peregrine Endoscope
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Endoscope Followed by Peregrine Drivable ENT Scope: Participants with prior endoscopic sinus surgery (EES) scheduled for nasal endoscopy who are receiving an endoscopy with the standard 30° 4mm endoscope followed by an endoscopy with the Peregrine Drivable ENT Scope.
Arm/Group | Standard Endoscope Followed by Peregrine Drivable ENT Scope
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.83 (17.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Visualization Success of Maxillary Sinus Anatomy
Description: The ability of each endoscope type to visualize the maxillary sinus anatomy (ostium, floor, lateral recess, anterior wall) was assessed as being a success or failure.
Time Frame: Day 1 (after each endoscopy)
Measure: Count of Participants; unit: Participants
Groups:
- Peregrine Drivable ENT Scope: Participants receiving an endoscopy with the Peregrine Drivable ENT scope.
- Standard 30° 4mm Endoscope: Participants receiving an endoscopy with the standard 30° 4mm endoscope.
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
Participants
  Left Ostium | 6 | 6
  Right Ostium | 6 | 6
  Left Floor | 6 | 1
  Right Floor | 4 | 0
  Left Lateral Recess | 6 | 1
  Right Lateral Recess | 5 | 1
  Left Anterior Wall | 6 | 0
  Right Anterior Wall | 4 | 0

2. Primary Outcome: Number of Participants With Visualization Success of Frontal Sinus Anatomy
Description: The ability of each endoscope type to visualize the frontal sinus anatomy (ostium, posterior table, anterior table, lateral recess) was assessed as being a success or failure.
Time Frame: Day 1 (after each endoscopy)
Measure: Count of Participants; unit: Participants
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
Participants
  Left Ostium | 6 | 6
  Right Ostium | 6 | 6
  Left Posterior Table | 4 | 3
  Right Posterior Table | 3 | 3
  Left Anterior Table | 4 | 2
  Right Anterior Table | 3 | 2
  Left Lateral Recess | 2 | 0
  Right Lateral Recess | 1 | 0

3. Primary Outcome: Number of Participants With Visualization Success of Sphenoid Sinus Anatomy
Description: The ability of each endoscope type to visualize the sphenoid sinus anatomy (ostium, sella, floor, lateral aspect) was assessed as being a success or failure.
Time Frame: Day 1 (after each endoscopy)
Measure: Count of Participants; unit: Participants
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
Participants
  Left Ostium | 6 | 5
  Right Ostium | 6 | 6
  Left Sella | 4 | 5
  Right Sella | 4 | 5
  Left Floor | 3 | 3
  Right Floor | 5 | 3
  Left Lateral Aspect | 4 | 2
  Right Lateral Aspect | 5 | 2

4. Secondary Outcome: Number of Participants With Adequate or Inadequate Image Quality From Peregrine Endoscopy
Description: Image quality will be assessed through a yes/no statement, reported by physicians, regarding the adequacy of the Peregrine image quality for making clinical decisions in the office setting.
Time Frame: Day 1 (after each endoscopy)
Measure: Count of Participants; unit: Participants
Arm/Group | Peregrine Drivable ENT Scope
Number analyzed (Participants) | 6
Participants
  Adequate image quality | 4
  Inadequate image quality | 2

5. Secondary Outcome: Visual Analogue Scale (VAS) Tolerability Score
Description: Participant tolerability was evaluated through validated VAS for both endoscopies. Scores range from 1 to 10, where 1 = highly tolerable and 10 = not tolerable.
Time Frame: Day 1 (after each endoscopy)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
score on a scale | 1.98 (1.72) | 2.52 (3.66)

6. Secondary Outcome: VAS Pain Score
Description: Participant pain was evaluated through validated VAS for both endoscopies. Scores range from 1 to 10, where 1 = no pain and 10 = pain as bad as it could be.
Time Frame: Day 1 (after each endoscopy)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
score on a scale | 3.75 (1.79) | 4.13 (3.5)

7. Secondary Outcome: Impact on Clinical Workflow
Description: The impact on clinical workflow of visual information obtained by each endoscope procedures was rated by physicians on a 5-point scale where 1 = worst and 5 = best.
Time Frame: Day 1 (after each endoscopy)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
score on a scale | 3 (1.55) | 5 (0)

8. Secondary Outcome: Ease of Use
Description: The ease of use of each endoscope procedure was rated by physicians on a 5-point scale where 1 = worst and 5 = best.
Time Frame: Day 1 (after each endoscopy)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
Number analyzed (Participants) | 6 | 6
score on a scale | 2.67 (1.37) | 5 (0)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the start of the procedure through the follow-up telephone call which occurred up to 2 weeks and 3 days after the procedure.
Arm/Group | Peregrine Drivable ENT Scope | Standard 30° 4mm Endoscope
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT04096482/Prot_SAP_000.pdf